CLINICAL TRIAL: NCT02052752
Title: A Randomized, Double-blinded Study to Evaluate the Ability of an Acne Treatment Product to Produce Visible Improvements in Acne Lesions Over a 5 Day Period of Once-daily Use
Brief Title: A Five Day Clinical Study to Examine the Effects of a Benzoyl Peroxide Treatment on Facial Acne Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201244; RH02060 (Other: GSK)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases | interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): Test product contained 3% benzoyl peroxide in the form of a gel. It was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Interventions: Drug: 3% Benzoyl Peroxide
- Vehicle gel (Active Comparator): The vehicle gel was similar to the test product except that it did not contain 3% benzoyl peroxide. The vehicle gel served as the negative control and was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Interventions: Drug: 3% Benzoyl Peroxide Placebo
- Positive control (Placebo Comparator): A commercial product containing 2% salicylic acid that reportedly improves acne lesions was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Interventions: Drug: Neutrogena Rapid Clear®

INTERVENTIONS:
Drug: 3% Benzoyl Peroxide — Test product contained 3% benzoyl peroxide in the form of a gel. It was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Arms: Test Product
Drug: 3% Benzoyl Peroxide Placebo — The vehicle gel was similar to the test product except that it did not contain 3% benzoyl peroxide. The vehicle gel served as the negative control and was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Arms: Vehicle gel
Drug: Neutrogena Rapid Clear® — A commercial product containing 2% salicylic acid that reportedly improves acne lesions was applied on participant's face once-daily at approximately the same time on Days 0, 1, 2 and 3.
  Arms: Positive control

SUMMARY:
5 Day study to assess how quickly a topical acne product begins to work.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
2. Fitzpatrick Skin Type I - V.
3. Male or female aged from 12 to 45 years, inclusive, at time of consent.
4. Mild to moderate facial acne vulgaris as determined by the Investigator, with a minimum of 10 inflammatory lesions (papules plus pustules, including nasal lesions) and a minimum of 10 non-inflammatory lesions (open and closed comedones, including nasal lesions).
5. Three appropriate and evaluable target lesions, as judged by the Investigator.
6. Able to complete the study and to comply with study instructions.
7. Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods include the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
   * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female participant has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Participants with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermicide is acceptable.
   * Women who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study.

Exclusion Criteria:

1. Has any nodulocystic lesions at the baseline evaluation.
2. Female who is pregnant, trying to become pregnant, or breastfeeding.
3. Has active or chronic skin allergies.
4. Has a history of acute or chronic disease that might interfere with or increase the risk of study participation.
5. Had skin cancer treatment in preceding 12 months.
6. Has damaged skin on facial areas (e.g., sunburn, tattoo, or scar).
7. Had any medical procedure (e.g., laser resurfacing, chemical peel, or plastic surgery) on facial areas in preceding 12 months.
8. Had any cosmetic procedure (e.g., microdermabrasion) on facial areas within 8 weeks of the baseline visit.
9. Has any dermatological disorder that in the opinion of the Investigator may interfere with the accurate evaluation of the participant's facial appearance.
10. Received any investigational drug or procedure within 28 days of study day 1 or is scheduled to receive an investigational drug (other than the study products) or procedure during the study.
11. Currently using any medication that in the opinion of the Investigator may affect the evaluation of the study products or place the participant at undue risk.
12. Has a history of known or suspected intolerance to any of the ingredients of the study products (i.e., benzoyl peroxide).
13. Considered unable or unlikely to attend the necessary visits.
14. Has used non-steroidal anti-inflammatory drugs for the treatment of acne or for treatment durations longer than 7 days for any condition.
15. Uses oil-based sunscreens or sunscreens containing active ingredients that may have an effect on acne.
16. Has received treatment with estrogens (including oral, implanted, and topical contraceptives), androgens, or anti-androgenic agents for 12 weeks or less immediately prior to starting application of the study product. Participants who have been treated with estrogens, as described above, androgens, or anti-androgenic agents for more than 12 consecutive weeks prior to starting application of the study product are allowed to enroll as long as they do not expect to change dose, drug, or discontinue use during the study.
17. Has used topical antibiotics on the face or use of systemic antibiotics within the previous 2 weeks.
18. Has used topical anti-acne medications (e.g., BPO, azelaic acid, resorcinol, salicylates) within the previous 2 weeks.
19. Has used topical corticosteroids on the face or systemic corticosteroids within the previous 4 weeks. Use of inhaled, intra-articular or intra-lesional steroids other than for facial acne is acceptable.
20. Has used systemic retinoids within the previous 6 months or topical retinoids within the previous 6 weeks.
21. Uses abradants, facials, peels containing glycolic or other acids; masks, washes or soaps containing BPO, salicylic acid, or sulfacetamide sodium; non-mild facial cleansers, or moisturizers that contain retinol, salicylic acid or α- or β-hydroxy acids.
22. Uses medications known to exacerbate acne (e.g., mega-doses of vitamin D [>2000 IU/day] and vitamin B12 [>1 mg/day]; systemic steroids; androgens; haloperidol; halogens such as iodide and bromide; lithium; hydantoin; and phenobarbital).
23. Has had any facial procedure (e.g., blue light, chemical or laser peel, microdermabrasion) performed by any practitioner within 4 weeks before the study started or during the course of the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a clinical site in USA
Pre-assignment Details: A total of 90 participants were randomized across the three treatment groups.
Period: Overall Study
Arm/Group | Test Product | Vehicle Gel | Positive Control
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Vehicle Gel | Positive Control | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.1 (9.90) | 20.3 (7.47) | 17.8 (6.22) | 20.1 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 (60.0) | 17 (56.7) | 12 (40.0) | 47
  Male | 12 (40.0) | 13 (43.3) | 18 (60.0) | 43

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Percentage Change in Acne Lesion Swelling (Height) of the Target Lesion for 3% Benzoyl Peroxide (BPO) Gel Test Product Relative to the Vehicle Gel After 4 Once-daily Applications.
Description: The Investigator assessed and score each target lesion's swelling (elevation), elevation scores were the actual dimensions, i.e. the value in millimeters at the lesion's highest points. Percent change in height of all three target lesions were calculated and averaged for each participant. The average lesion height at baseline was calculated for each participant. An analysis of covariance (ANCOVA) was performed with average percentage change in target lesion height as the response variable, treatment group (3% BPO or vehicle) as a main effect, and average baseline target lesion height as a covariate. A greater reduction in the percentage change in height of the target lesions indicated a better outcome measure
Time Frame: Baseline to Day 4
Population: The analysis population consists of the intent-to-treat (ITT) population. The ITT analysis set comprised of all participants who were randomized and received at least 1 application of study product and had baseline assessment.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Percentage change | -57.42 (6.229) | -47.89 (6.237) | -53.07 (6.233)
Statistical Analysis 1: Comparison: Test Product vs Vehicle Gel; The ANCOVA results for the primary endpoint with treatment group as a main effect and average baseline value as a covariate showed no statistically significant differences in the percentage change from baseline in swelling of the target lesions between the 3% BPO group and the vehicle control group at Day 4 for the ITT population; Test type: Superiority or Other; p = 0.283, ANCOVA

2. Secondary Outcome: To Assess the Percentage Change in Acne Lesion Swelling (Height) for the 3% Benzoyl Peroxide Gel Test Product and Positive Control Relative to the Vehicle Gel.
Description: The Investigator assessed and score each target lesion's swelling (elevation), elevation scores were the actual dimensions, i.e. the value in millimeters at the lesion's highest points. Percent change in height of all three target lesions were calculated and averaged for each participant. The average lesion height at baseline was calculated for each participant
Time Frame: Baseline to 2 hours, 4 hours, Day 1, Day 2 and Day 4
Population: The analysis population consists of the ITT population. The ITT analysis set comprised of all participants who were randomized and received at least 1 application of study product and had baseline assessment.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Percentage change
  From baseline to hour 2 | -3.24 (8.726) | -4.65 (10.558) | -4.57 (10.754)
  From baseline to hour 4 | -6.02 (9.172) | -7.01 (11.525) | -5.94 (11.774)
  From baseline to day 1 | -21.42 (25.578) | -22.07 (19.688) | -20.22 (25.711)
  From baseline to day 2 | -40.30 (34.011) | -37.03 (28.968) | -42.94 (31.121)
  From baseline to day 4 | -57.22 (36.372) | -48.60 (34.585) | -52.57 (33.580)

3. Secondary Outcome: To Assess the Change in Acne Lesion Redness (Erythema) for the 3% BPO Gel Test Product and Positive Control Relative to the Vehicle Gel.
Description: The investigator assessed the erythema of the target lesion according to the following scale and tabulated the responses: 0=none, 1=minimal, 2=mild, 3=-moderate, 4=severe.
Time Frame: Baseline to 2 hours, 4 hours, Day 1, Day 2, and Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale
  Change from baseline to hour 2 | -0.04 (0.190) | -0.02 (0.122) | -0.03 (0.221)
  Change from baseline to hour 4 | -0.12 (0.283) | -0.06 (0.304) | -0.10 (0.279)
  Change from baseline to day 1 | -0.62 (0.811) | -0.56 (0.639) | -0.73 (0.851)
  Change from baseline to day 2 | -1.26 (1.225) | -1.02 (0.967) | -1.36 (1.168)
  Change from baseline to day 4 | -1.83 (1.228) | -1.39 (1.247) | -1.84 (1.303)

4. Secondary Outcome: To Assess the Percentage Change in Acne Lesion Diameter (Size) for the 3% BPO Gel Test Product and Positive Control Relative to the Vehicle Gel.
Description: The Investigator assessed and score each target lesion's diameter (size). Diameter scores were the actual dimensions, i.e. the value in millimeters at the lesion's widest or highest points.
Time Frame: Baseline to 2 hours, 4 hours, Day 1, Day 2, and Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Percentage change
  From baseline to hour 2 | -0.46 (10.920) | -1.33 (7.274) | -0.33 (7.112)
  From baseline to hour 4 | -0.74 (9.397) | -0.22 (10.666) | -0.63 (9.244)
  From baseline to day 1 | -12.46 (27.993) | -12.83 (20.836) | -11.93 (22.049)
  From baseline to day 2 | -30.98 (38.935) | -29.81 (36.983) | -37.83 (32.315)
  From baseline to day 4 | -52.56 (39.058) | -38.78 (44.7000) | -44.78 (35.933)

5. Secondary Outcome: To Assess the Change in Facial Skin Clarity for the 3% BPO Gel Test Product and Positive Control Relative to the Vehicle Gel
Description: The Skin clarity was measured using the following scale; 0 Very Clear; 1 Clear; 2 Dull; 3 Very Dull; 4 Unclear. The responses were then tabulated
Time Frame: Baseline to 2 hours, 4 hours, Day 1, Day 2, and Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale
  Baseline to hour 2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Baseline to hour 4 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Baseline to day 1 | -0.2 (0.43) | -0.2 (0.38) | -0.3 (0.48)
  Baseline to day 2 | -0.8 (0.81) | -0.5 (0.51) | -0.7 (0.84)
  Baseline to day 4 | -1.2 (0.90) | -0.7 (0.79) | -1.0 (0.98)

6. Secondary Outcome: To Assess the Change in Perceptions of the Overall Appearance of Their Skin for the 3% BPO Gel Test Product and Positive Control Relative to the Vehicle Gel
Description: The participants were asked to rate the overall appearance of their facial skin as; 1= Very Dissatisfied; 2= Slightly Dissatisfied; 3= Neither Satisfied nor Dissatisfied; 4= Slightly Satisfied; 5= Very Satisfied. The responses were then tabulated.
Time Frame: Baseline to 2 hours, 4 hours, Day 1, Day 2, and Day 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test Product | Vehicle Gel | Positive Control
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale
  Change from baseline to hour 2 | 0.3 (0.84) | 0.1 (0.82) | 0.3 (0.71)
  Change from baseline to hour 4 | 0.4 (0.93) | 0.3 (0.99) | 0.4 (1.07)
  Change from baseline to day 1 | 0.3 (0.92) | 0.3 (1.03) | 0.4 (1.13)
  Change from baseline to day 2 | 0.5 (1.14) | 0.6 (1.03) | 0.7 (1.24)
  Change from baseline to day 4 | 0.9 (1.03) | 0.8 (1.30) | 0.8 (1.32)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Test Product | Vehicle Gel | Positive Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.